CLINICAL TRIAL: NCT04764942
Title: Phase 1/2 Trial of Selinexor in Combination With Pomalidomide and Dexamethasone ± Carfilzomib for Patients With Proteasome-Inhibitor and Immunomodulatory Drug Refractory Multiple Myeloma (SCOPE)
Brief Title: Selinexor, Pomalidomide, and Dexamethasone With or Without Carfilzomib for the Treatment of Patients With Relapsed Refractory Multiple Myeloma, The SCOPE Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1882; NCI-2021-01268 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; pomalidomide; selinexor; X-Rays; Phantoms, Imaging; Magnetic Resonance Spectroscopy; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (selinexor, dexamethasone, carfilzomib, carfilzomib) (Experimental): Patients receive selinexor PO and dexamethasone PO on days 1, 8 15, and 22, carfilzomib IV on days 1, 8, and 15, and pomalidomide PO on days 1-21. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT or CT and bone marrow biopsy and aspiration during screening and on the trial. Patients may optionally undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Pomalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selinexor; Procedure: X-Ray Imaging; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection
- Arm B (selinexor, dexamethasone, pomalidomide) (Experimental): Patients receive selinexor PO and dexamethasone PO on days 1, 8, 15, and 22, and pomalidomide PO on days 1-21. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT or CT and bone marrow biopsy and aspiration during screening and on the trial. Patients may optionally undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Dexamethasone; Drug: Pomalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selinexor; Procedure: X-Ray Imaging; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR-171
  Arms: Arm A (selinexor, dexamethasone, carfilzomib, carfilzomib)
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Static X-Ray; X-Ray
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; CT; CT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; Proton magnetic resonance spectroscopic imaging
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection; Blood Sample Collection

SUMMARY:
This phase I/II trial identifies the best dose and side effects of selinexor, and how well it works when given in combination with pomalidomide and dexamethasone with or without carfilzomib in treating patients with multiple myeloma that has come back (relapsed) and does not respond to treatment with proteasome inhibitors and immunomodulatory drugs (refractory). Selinexor is an oral agent that blocks a protein called Exportin 1 (XPO1 or CRM1) that is abundant in a wide variety of cancers, including multiple myeloma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Pomalidomide may stop the growth of blood vessels, stimulate the immune system, and kill cancer cells. Anti-inflammatory drugs, such as dexamethasone may lower the body's immune response and are used with other drugs in the treatment of some types of cancer. The addition of selinexor may allow better control of relapsed refractory multiple myeloma than is possible with pomalidomide and dexamethasone with or without carfilzomib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of selinexor in combination with carfilzomib, pomalidomide and dexamethasone (SKPd) in patients with relapsed refractory multiple myeloma (RRMM). (Arm A) II. To determine the efficacy of fixed-dose selinexor in combination with low-dose pomalidomide and dexamethasone (SPd) in patients with RRMM as measured by the overall response rate (ORR) per the International Myeloma Working Group (IMWG) criteria. (Arm B)

SECONDARY OBJECTIVES:

I. To evaluate the preliminary efficacy of SKPd in relapsed/refractory multiple myeloma, as measured by the overall response rate (ORR) per International Myeloma Working Group (IMWG) criteria and the duration of response (DOR). (Arm A) II. To evaluate clinical benefit rate (CBR), duration of response, progression-free survival, overall survival, and the safety profile of SPd. (Arm B)

EXPLORATORY OBJECTIVES:

I. To estimate clinical activity in different risk groups by cytogenetics. II. To assess minimal residual disease by flow cytometry in patients achieving complete response (CR) and compare the outcomes of patients who are serum mass-fix (mass spectrometry-based methodology available at Mayo Clinic) negative only versus those who have no evidence of disease by mass fix and flow-cytometry-based minimal residual disease (MRD).

III. To assess overall health-related quality of life, as measured by the global health domain of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire and Quality of Life Questionnaire-Multiple Myeloma 20 (QLQ-MY20).

IV. To evaluate patient reported outcomes using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (Patient Reported Outcomes Version of Common Terminology Criteria for Adverse Events [PRO-CTCAE]).

V. To stratify patients in arm A based on quadruple/penta-refractory status and to assess the impact of this stratification on patient outcomes.

VI. To stratify patients in arm B based on their dual-refractory status and to assess the impact of this stratification on patient outcomes.

OUTLINE: Patients with >= 3 prior lines of therapy are assigned to Arm A, while patients with 1-2 prior lines of therapy are assigned to Arm B. Arm A is a phase I dose-escalation study of selinexor and carfilzomib, with fixed-dose dexamethasone and pomalidomide followed by a dose-expansion study. Arm B is a phase II fixed-dose study of selinexor, dexamethasone, and pomalidomide.

ARM A: Patients receive selinexor orally (PO) and dexamethasone PO on days 1, 8 15, and 22, carfilzomib intravenously (IV) on days 1, 8, and 15, and pomalidomide PO on days 1-21. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo x-ray imaging during screening. Patients also undergo positron emission tomography/computed tomography (PET/CT) or CT and bone marrow biopsy and aspiration during screening and on the trial. Patients may optionally undergo blood sample collection during screening and on the trial.

ARM B: Patients receive selinexor PO and dexamethasone PO on days 1, 8, 15, and 22, and pomalidomide PO on days 1-21. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo x-ray imaging during screening. Patients also undergo PET/CT or CT and bone marrow biopsy and aspiration during screening and on the trial. Patients may optionally undergo blood sample collection during screening and on the trial.

After completion of study treatment, patients are followed up at 30 days, then every 3 months until progressive disease (PD) or subsequent treatment, then every 6 months until 3 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of RRMM with progressive disease at study entry as per the International Myeloma Working Group (IMWG) uniform criteria
* Measurable disease by IMWG criteria as defined by at least one of the following:

  * Serum M-protein >= 0.5 g/dL
  * Urine M-protein >= 200 mg in a 24-hour collection
  * Serum free light chain level >= 10 mg/dL provided the free light chain ratio is abnormal
  * For patients with extramedullary measurable disease (EMD) by CT or MRI or the CT portion of the PET/CT: Must have at least one lesion that has a single diameter of >= 2 cm. Skin lesions can be used if the area is >= 2cm in at least one diameter and measured with a ruler
  * Bone marrow plasma cells >= 30%
  * Patients with IgA myeloma in whom serum protein electrophoresis is deemed unreliable, due to co-migration of normal serum proteins with the para protein in the beta region, may be considered eligible as long as total serum IgA level is elevated above normal range
* Prior treatment:

  * Arm A: At least one of the following must be true: (1) Subjects must have been previously treated with at least 3 prior lines of therapy, including a proteasome inhibitor and an immunomodulatory drug (IMiD) (2) Subjects who are refractory to carfilzomib and/or pomalidomide may enroll in Arm A using the quadruplet regimen, SKPd, provided carfilzomib, pomalidomide and dexamethasone (KPd) triplet is not the most recent line of prior therapy and that they have been previously treated with at least 3 prior lines of therapy, including a proteasome inhibitor and an IMiD. Carfilzomib/Pomalidomide refractory status is defined by the IMWG criteria: disease that is nonresponsive (stable disease [SD] or progressive disease [PD]) while on therapy, or progresses within 60 days of last therapy in patients who have achieved minimal response (MR) or better at some point previously before then progressing in their disease course.
  * Arm B: Subjects must have progressive disease and been exposed to up to 2 prior lines of therapy, including a proteasome inhibitor and lenalidomide
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study) and ability to adhere with the study visit schedule and other protocol procedures
* Willingness to provide mandatory tissue specimens for correlative research
* Willingness to use fixed-duration therapy (up to 18 cycles) for relapsed refractory multiple myeloma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 15 mL/min (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/uL(without growth factor support for >= 7 days ( obtained =< 14 days prior to registration)
* Un-transfused Platelet count >= 100,000/uL (without platelet transfusion for >= 14 days) for SKPd and >= 100,000 (without platelet transfusion for >= 7 days) for SPd is permitted. Additionally, for both Arms A and B platelet count of >= 75,000/uL is permitted if thrombocytopenia is deemed by the investigator to be secondary to severe bone marrow infiltration (>= 50%) by myeloma as determined
* Hemoglobin >= 8.0 g/dL Note: Screening hemoglobin should be independent of red blood cell transfusion for at least 3 days prior to screening
* Total bilirubin =< 2.0 x upper limit of normal (ULN). Note: Patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN

  * Note: If patient is receiving warfarin and INR should be within 2-3
* Negative serum pregnancy test done =<7 days prior to registration, for persons of childbearing potential only
* Willingness to follow strict birth control measures as suggested by the study: Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for 28 days prior to starting pomalidomide, during the course of the study, during any dose interruptions, and through 30 days after last dose of pomalidomide and carfilzomib. Female subjects of child bearing potential are those who 1) have achieved menarche at some point, 2) have not undergone a hysterectomy or bilateral oophorectomy or 3) have not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Male subjects must agree to practice abstinence or use an effective barrier method of contraception starting with the first dose of carfilzomib or pomalidomide through 6 months after last dose of pomalidomide and carfilzomib if sexually active with a female of childbearing potential. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Other acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. All subjects must agree to follow the local requirements for pomalidomide counseling, pregnancy testing, and birth control; and be willing and able to comply with the local requirements (for example, periodic pregnancy tests, safety labs, etc.)
* Willingness to follow the requirements of the Pomalyst Risk Evaluation and Mitigation Strategy (REMS) program
* Able to swallow capsules and able to take and tolerate oral medications on a continuous basis

Exclusion Criteria:

* History of myocardial infarction =< 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias. Unstable angina within 4 months prior to randomization, New York Heart Association (NYHA) class III or IV heart failure, left ventricular ejection fraction (LVEF) < 40%, uncontrolled angina, corrected QT (QTc) interval >= 470 msec, History of severe coronary artery disease, severe uncontrolled ventricular arrhythmias including uncontrolled chronic atrial fibrillation/atrial flutter, history of torsades de pointe, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment.

EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 1 month since completion of prior treatment

* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals =< 14 days prior to registration; patients with controlled infection or on prophylactic antibiotics are permitted in the study
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Patients known to be human immunodeficiency virus (HIV) positive and/or currently receiving antiretroviral therapy
* Currently receiving any other investigational agent which would be considered as a treatment for RRMM
* Non investigational radiation, chemotherapy, or immunotherapy or any other anticancer therapy =< 14 days or five half-lives, whichever is shorter prior to registration. Note: (localized radiation to a single site =< 7 days prior to registration is allowed)
* Participation in an investigational anti-cancer study =< 21 days or five half-lives whichever is shorter prior to registration
* Major Surgery =< 21 days prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Other active malignancy =< 5 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix that has undergone potentially curative therapy. NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Uncontrolled hypertension or uncontrolled diabetes =< 14 days prior to registration
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) ribonucleic acid (RNA) or hepatitis B surface antigen (HBsAg) [hepatitis B virus (HBV) surface antigen]
* Significant neuropathy (grades 3-4, or grade 2 with pain) =< 14 days prior to registration
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis =< 14 days prior to registration
* Patients with coagulation problems and active bleeding in the last month (e.g, peptic ulcer, epistaxis, spontaneous bleeding)
* Subjects with smoldering multiple myeloma (SMM), monoclonal gammopathy of undetermined significance (MGUS) or Waldenström's macroglobulinemia or AL amyloidosis
* History of repeated infections, hyperviscosity or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Has a known history of immunosuppression or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy =< 7 days prior registration. The use of physiologic doses of corticosteroids may be approved after consultation with the study chair

  * Note: A short course of 40 mg dexamethasone (=< 4 days) or equivalent for emergency use is allowed after previous consultation with the study chair. In these cases, baseline m-protein values from serum and urine should be obtained before the short steroid course and be repeated prior to study drugs administration on cycle 1 day 1
* Treatment with plasmapheresis =< 28 days prior to registration
* Known hypersensitivity to thalidomide, lenalidomide or dexamethasone
* Unable or unwilling to undergo thromboembolic prophylaxis including, as clinically indicated, aspirin, Coumadin (warfarin) or low-molecular weight heparin
* Evidence of active, non-infectious pneumonitis
* Received a live vaccine =< 30 days prior to registration
* Pomalidomide and carfilzomib (for arm A) or pomalidomide (for Arm B) commercially unavailable to the patient
* Prior exposure to Selinexor
* Pregnant persons

  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception (applies to both male and female participants as written)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of selinexor in combination with carfilzomib, pomalidomide and dexamethasone (Phase I) | Up to 30 days after completion of treatment
  A standard 3+3 phase I design will be utilized. Three patients will be treated at each dose level and observed for a minimum of four weeks (i.e. one full cycle) before new patients are treated. Doses will not be escalated in any individual patient.
Proportion of patients who achieve a confirmed response with selinexor in combination with pomalidomide and dexamethasone (Phase 2) | Up to 3 years
  A confirmed response is defined as an stringent complete response (sCR), complete response (CR), very good [partial response (VGPR), or partial response (PR) noted as the objective status on two consecutive evaluations. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Duration of response | Up to 3 years
  Defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be an sCR, CR, VGPR, or PR to the earliest date progression or relapse is documented.
Clinical benefit rate | Up to 3 years
  Will be estimated by the number of patients with an sCR, CR, VGPR, PR, or MR noted as the objective status on two consecutive evaluations divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Overall survival | From registration to death due to any cause, assessed up to 3 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier
Progression-free survival | From registration to the earliest date of documentation of disease progression, relapse, or death due to any cause, assessed up to 3 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
  Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.

OTHER OUTCOMES:
Relationship between risk groups | Up to 3 years
  Patients will be categorized into different risk groups by cytogenetics and gene expression profiling. The relationship between risk groups and outcomes (confirmed response and progression-free survival) will be evaluated using Kruskal Wallace and log rank tests.
Minimal residual disease (MRD) | Up to 3 years
  Will be assessed on bone marrow aspirate in all patients achieving sCR or CR. The proportion of patients who achieve MRD negative status will be estimated by the number of patients who are MRD negative divided by the total number of evaluable patients who achieve an sCR or CR. Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Overall health-related quality of life | Up to 18 cycles (each cycle is 28 days)
  Will be assessed through patient self-reported instruments including the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 and Multiple Myeloma-20 instruments. High scores for the both global and functional domains indicate higher quality of life or functioning, while high scores on the symptom scales represent higher levels of symptomatology or problems.
Patient reported outcomes (PRO) | Up to 3 years
  The PRO-Common Terminology Criteria for Adverse Events (CTCAE) will be incorporated to provide a better understanding of patient-reported symptomatic toxicity. PRO-CTCAE scores range from 0-4, with corresponding response choices for frequency (never / rarely / occasionally / frequently / almost constantly), for severity (none / mild
  / moderate / severe / very severe) and interference (not at all / a little bit / somewhat / quite a bit / very much). The scores for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. PRO-CTCAE data will be summarized descriptively as the number (%) of patients reporting each grade for individual items, and all available attribute items, will be included for each of the reported symptoms. The analyses will be exploratory and descriptive, and no statistical comparisons will be conducted. The relationship between refractory status and patient outcome will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kapoor, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials